CLINICAL TRIAL: NCT03206606
Title: Evaluation of a Mobile Application to Facilitate the Interpretation of the Spirometry Test by Family Physicians and Family Medicine Residents: Impact on Prescription and Interpretation of This Test
Brief Title: Evaluation of a Mobile Application to Facilitate the Interpretation of Spirometry by Family Physicians and Residents
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, Pneumologist, Laval University
Other Study IDs: SPIRO-MD Residents
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: COPD; Spirometry; Mobile Application
Keywords: COPD; Spirometry; Mobile application
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Primary care physicians and residents in family medicine of family medicine units affiliated with Laval University.
- Experimental Group: Primary care physicians and residents in family medicine of family medicine units affiliated with Laval University that will use the mobile application SPIRO(c) for a period of four months.
  Interventions: Device: SPIRO

INTERVENTIONS:
Device: SPIRO — Participants in the Experimental Group will be asked to use SPIRO mobile application during a period of 4 months.
  Groups: Experimental Group

SUMMARY:
Problematic: Spirometry is used to objectify the obstructive syndrome defining chronic obstructive pulmonary disease (COPD). However, this test remains underused in the primary care. The tools available for its interpretation are little used and the existence of several decision algorithms can create confusion during the diagnosis.

Principal objective: To evaluate the impact of a mobile application (SPIRO©) on medical practice (interpretation and prescription of spirometry) of family physicians and family medicine residents working in family medicine units (FMU) in Quebec affiliated with Laval University.

Secondary objective : To evaluate the usability of SPIRO© among family physicians and residents in family medicine working in FMU in Quebec affiliated with Laval University.

Methods: This is a pre-post clinical trial with control group. Participants (family MD and family medicine residents) will be recruited from the various FMU affiliated with Laval University. Participants working in the FMU in the experimental group will be able to use the SPIRO® mobile application to facilitate interpretation of the spirometry test results while participants in the control group will not have access to it during the study. The basic characteristics of the participants and various behavioral parameters based on the theory of planned behavior concerning the interpretation and prescription of spirometry test will be measured. Data from the control group will be collected before those in the experimental group at the time the application is not yet available, which will minimize contamination between groups. The data will be collected with questionnaires delivered in person to the participants before the intervention (T0 time) and then four months later (T1 time) during their team or research meeting. Participants will be recruited in eight of the 12 Quebec FMU affiliated with Laval University, who will be randomly assigned to two equal groups: control and experimental. The intervention will consist in sending the SPIRO© mobile application to participants in the experimental group who will use it for a period of four months.

DETAILED DESCRIPTION:
Hypothesis : The investigators hypothesize that the use of the SPIRO© application will increase the skills and confidence of family physicians and family medicine residents in prescribing and interpreting spirometry compared to the control group.

The project will be conducted in the following six major steps: 1) Collection of socio-demographic and behavioral characteristics of participants using sections A, B, C and D of the NAPI questionnaire in the control group; 2) Intervention in the control group (they will continue their daily medical practice without being subject to any intervention by our research team), for a period of 4 months; 3) Measurement of behavioral changes in the control group using Sections B, C, D and E of the NAPI questionnaire 4 months after the start of the study; 4) Collection of socio-demographic and behavioral data from participants in the experimental group using sections A, B, C and D of the NAPI questionnaire; 5) E-mail distribution of the application and use of the application by participants in the experimental group for a period of four months, 6) Measurement of behavioral changes in the experimental group after the use of the application, Using sections B, C, D and E of the NAPI questionnaire as well as a questionnaire on the application SPIRO© (SPIRO questionnaire) which will evaluate the usability of this one.

The study has been approved by the research ethic board of the Health and Social Services Center of the old capital - attached to the Integrated Center for Health and Social Services of the National Capital.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to be primary care physicians or residents in family medicine of 18 years old or more working in one of the 12 family medicine units in Quebec affiliated with Laval University.

Exclusion Criteria:

* Health professionals not practicing family medicine and residents of other specialties will not be eligible. Individuals who participated in the development of the " subjective Norms, Attitudes, Perceived behavioral control, Intentions (NAPI) " questionnaires (apparent validation) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care physicians and residents in family medicine of 18 years old or more working in one of the 12 family medicine units in Quebec affiliated with Laval University.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Beliefs about capabilities - interpretation | six weeks
  The beliefs about the capabilities of primary care physicians and residents in family medicine regarding interpretation of spirometry.

SECONDARY OUTCOMES:
Beliefs about consequences - prescription | six weeks
  The beliefs about the consequences of primary care physicians and residents in family medicine regarding prescription of spirometry.
Beliefs about consequences - interpretation | six weeks
  The beliefs about the consequences of primary care physicians and residents in family medicine regarding interpretation of spirometry.
Beliefs about consequences - use of a mobile application | six weeks
  The beliefs about the consequences of primary care physicians and residents in family medicine regarding the use of a mobile application to interpret spirometry.
Moral norms - prescription | six weeks
  The beliefs about the moral norms of primary care physicians and residents in family medicine regarding prescription of spirometry.
Moral norms - interpretation | six weeks
  The beliefs about the moral norms of primary care physicians and residents in family medicine regarding interpretation of spirometry.
Moral norms - use of a mobile application | six weeks
  The beliefs about the moral norms of primary care physicians and residents in family medicine regarding the use of a mobile application to interpret spirometry.
Intentions - prescription | six weeks
  The beliefs about the intentions of primary care physicians and residents in family medicine regarding prescription of spirometry.
Intentions - interpretation | six weeks
  The beliefs about the intentions of primary care physicians and residents in family medicine regarding interpretation of spirometry.
Intentions - use of a mobile application | six weeks
  The beliefs about the intentions of primary care physicians and residents in family medicine regarding the use of a mobile application to interpret spirometry.
Social influence - prescription | six weeks
  The beliefs about the social influence of primary care physicians and residents in family medicine regarding prescription of spirometry.
Social influence - interpretation | six weeks
  The beliefs about the social influence of primary care physicians and residents in family medicine regarding interpretation of spirometry.
Social influence - use of a mobile application | six weeks
  The beliefs about the social influence of primary care physicians and residents in family medicine regarding the use of a mobile application to interpret spirometry.
Belief about capabilities - prescription | six weeks
  The beliefs about the belief about capabilities of primary care physicians and residents in family medicine regarding prescription of spirometry.
Belief about capabilities - use of a mobile application | six weeks
  The beliefs about the belief about capabilities of primary care physicians and residents in family medicine regarding the use of a mobile application to interpret spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Heart and Lung Institute
Locations (8):
- Canada (8):
  - UMF de Manicouagan, Baie-Comeau, Quebec
  - UMF de Gaspé, Gaspé, Quebec
  - UMF des Etchemins, Lac-Etchemin, Quebec
  - UMF de Lévis, Lévis, Quebec
  - Unité de médecine familiale - GMF Maizerets, Québec, Quebec
  - UMF Saint-François d'Assise, Québec, Quebec
  - Unité de médecine familiale Laval, Québec, Quebec
  - UMF de Trois-Pistoles, Trois Pistoles, Quebec

IPD SHARING:
Plan to Share IPD: Undecided